CLINICAL TRIAL: NCT05923437
Title: Effect of Chronobıologıcal Approach Feedıng Model on Cırcadıan Rhythm, Growth and Physıologıcal Parameters in Newborn: A Randomızed Controlled Study
Brief Title: The Effect of Chronobiologic Feeding Model on Circadian Rhythm in Newborns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Sibel Küçükoğlu, Professor, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SelcukUnı42
Record Dates: First submitted 2023-06-20; First posted 2023-06-28 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Breast Feeding, Exclusive; Hospitalization; Feeding Patterns
Keywords: Breast milk; Nutrition; Nursing; Chronobiology; Circadian rhythm; Sleep wake cycle; Newborn
MeSH Terms: conditions — Breast Feeding; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: The study will be conducted with a total of 40 newborns (intervention group=20, control group= 20). In order to prevent selection bias in the study, participants will be randomly assigned to the intervention and control groups and the "block randomization" method, one of the "fixed probability randomization" methods, will be used in randomization. Each of the intervention and control groups will be represented by one of the letters A and B. In the creation of the 4-block (2A, 2B); the assignment of 10 blocks from the total number of options determined using the "permutation" method will be carried out with the random numbers table tool on the www.random.org website.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Interventions Group (Experimental): Breast milk will be given to the newborns in the intervention group for 3 days in line with the "feeding model with a chronobiological approach", simultaneously with the mother's supply.
  Interventions: Other: Feeding model group with a chronobiological approach
- Control Group (No Intervention): Breast milk will be given to newborns in the control group according to the clinical routine and infants will be followed up for 3 days.

INTERVENTIONS:
Other: Feeding model group with a chronobiological approach — Breast milk will be given to the newborns in the intervention group for 3 days in line with the "feeding model with a chronobiologic approach" simultaneously with the provision from the mother, and the newborn will be ensured to receive breast milk in accordance with the day cycle. Within the scope of the study, firstly, mothers and nurses in the NICU will be informed about the study. Mothers will be asked to put the milk mothers express between 06:00-17:59 in the "daytime breast milk storage bag" and the milk mothers express between 18:00-05:59 in the "nighttime breast milk storage bag" and bring them to the unit. The brought breast milk will be prepared by the nurses by matching "day and night" milk according to the dates, with the first milk brought in priority, and the newborns will be fed by using the "time of day factor" (cycle so that the milk collected during the day will be given during the day and the milk expressed at night will be given at night).
  Arms: Experimental: Interventions Group

SUMMARY:
This study was planned to evaluate the effect of "feeding model with chronobiologic approach" on circadian rhythm, growth and physiologic parameters of newborns.

DETAILED DESCRIPTION:
The newborn period is a period when all babies need their basic needs to be met and all babies are very sensitive physiologically, neuro-biologically and psycho-emotionally, but the newborn period is also a very important period in the development of circadian rhythm. It is important to establish a healthy sleep pattern for the formation of the circadian rhythm and the continuation of the functions of all other systems, especially the central nervous system. Formation of circadian rhythm in newborns; It shows a better development in the first 3 months with the effect of environmental factors such as nutrition, light, mother-baby interaction. Breast milk is a nutrient for the growth and development of babies, in addition, breast milk plays an active role in the formation of the baby's circadian rhythm by transmitting information about the time of day to the babies through components such as hormones and immune elements. In cases where breastfeeding is not possible, it is thought that the delivery of expressed breast milk to the babies simultaneously with the "feeding model with a chronobiological approach" has important effects on the sleep-wake cycle and growth and development. In studies examining circadian rhythm in newborns in the world and in our country, the limited number of studies evaluating the relationship between circadian rhythm and breast milk draws attention and further studies are recommended. However, there is no published study evaluating the effect of simultaneous administration of breast milk to the infant in line with the "feeding model with chronobiologic approach" on circadian rhythm, growth and physiologic parameters of newborns.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 28-42 weeks
* Birth weight between 1500 and 4200 gr
* Hospitalization for at least 3 days
* Exclusive breastfeeding (oral/ enteral)
* Feeding at 3-hour intervals
* Stable health condition
* Spontaneous breathing

Exclusion Criteria:

* Babies fed outside of 3-hour intervals (hourly or two-hourly intervals)
* 5th minute apgar score below 4 at the time of delivery
* Resuscitation requirement
* Having a congenital anomaly
* Interventional intervention in the head region
* Central nervous system dysfunction
* Postpartum medical complications

Ages: 28 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Newborn Introductory Information Form | First measurement - Before the study (before randomization)
  The form prepared by the researcher in line with the literature (Galland et al., 2012; Huang et al., 2021; Caba-Flores et al., 2022) consists of questions including the obstetric characteristics of the infant such as gender, gestational-postnatal age, type of delivery, APGAR scores, birth weight, height, head circumference, and the current clinical status of the infant such as diet, comorbidity, and total number of hospitalization days. The questionnaire form was sent to 5 academicians specialized in Pediatric Nursing, their expert opinions were obtained, and the questionnaire form was finalized by making the necessary changes in line with their suggestions. Information about the newborns in the control and experimental groups was collected by the researcher through the "Newborn Introductory Information Form" before the study, hospital records of the newborn and the primary nurse through face-to-face interview method will be collected in about 5 minutes.
Newborn Growth and Physiologic Parameters Follow-up Chart | First measurement - up the end of the first day night and day measurements
  "Temperature (°C), Pulse Rate (min), Blood Pressure (mmHg), Respiratory Rate (min), O2 Saturation (mmHg) will be recorded for 3 days during the day-night cycle of the infants followed in both groups. Physiologic parameters will be measured 1 hour after the 2nd daytime feeding and 1 hour after the 2nd nighttime feeding (i.e. after the baby's 6th feeding). The amount of breast milk received by the infant (ml)" will be monitored for three days separately in the daytime (06:00-17:59) and nighttime (18:00-05:59) cycle. In addition, the infants will be followed up in terms of "Body Weight (g), Height (cm), Head circumference (cm), Persentile" values until the infants are discharged from the hospital and all these parameters will be recorded through the "Newborn Growth and Physiological Parameters Follow-up Chart" created by the researcher.
Newborn Circadian Rhythm Follow-up Chart | First measurement -up the end of the first day circadian rhythm measurements
  At the end of 3 days, the records of the duration of the babies' being in "Wakefulness, REM, N-REM / EVRE I, N-REM / EVRE II, N-REM / EVRE III, N-REM / EVRE III, N-REM / EVRE IV" measured by Bispectral Index (BIS) in 5-minute periods within a 24-hour time cycle will be taken from the BIS monitor records and entered into the "Newborn Circadian Rhythm Follow-up Chart" created by the researcher.

SECONDARY OUTCOMES:
Newborn Growth and Physiologic Parameters Follow-up Chart | Second measurement - up the end of the second day night and day measurements
  "Temperature (°C), Pulse Rate (min), Blood Pressure (mmHg), Respiratory Rate (min), O2 Saturation (mmHg) will be recorded for 3 days during the day-night cycle of the infants followed in both groups. Physiologic parameters will be measured 1 hour after the 2nd daytime feeding and 1 hour after the 2nd nighttime feeding (i.e. after the baby's 6th feeding). The amount of breast milk received by the infant (ml)" will be monitored for three days separately in the daytime (06:00-17:59) and nighttime (18:00-05:59) cycle. In addition, the infants will be followed up in terms of "Body Weight (g), Height (cm), Head circumference (cm), Persentile" values until the infants are discharged from the hospital and all these parameters will be recorded through the "Newborn Growth and Physiological Parameters Follow-up Chart" created by the researcher.
Newborn Circadian Rhythm Follow-up Chart | Second measurement - up the end of the second day circadian rhythm measurements
  At the end of 3 days, the records of the duration of the babies' being in "Wakefulness, REM, N-REM / EVRE I, N-REM / EVRE II, N-REM / EVRE III, N-REM / EVRE III, N-REM / EVRE IV" measured by Bispectral Index (BIS) in 5-minute periods within a 24-hour time cycle will be taken from the BIS monitor records and entered into the "Newborn Circadian Rhythm Follow-up Chart" created by the researcher.
Newborn Growth and Physiologic Parameters Follow-up Chart | Third measurement - up the end of the third day night and day measurements
  "Temperature (°C), Pulse Rate (min), Blood Pressure (mmHg), Respiratory Rate (min), O2 Saturation (mmHg) will be recorded for 3 days during the day-night cycle of the infants followed in both groups. Physiologic parameters will be measured 1 hour after the 2nd daytime feeding and 1 hour after the 2nd nighttime feeding (i.e. after the baby's 6th feeding). The amount of breast milk received by the infant (ml)" will be monitored for three days separately in the daytime (06:00-17:59) and nighttime (18:00-05:59) cycle. In addition, the infants will be followed up in terms of "Body Weight (g), Height (cm), Head circumference (cm), Persentile" values until the infants are discharged from the hospital and all these parameters will be recorded through the "Newborn Growth and Physiological Parameters Follow-up Chart" created by the researcher.
Newborn Circadian Rhythm Follow-up Chart | Third measurement - up the end of the third day circadian rhythm measurements
  At the end of 3 days, the records of the duration of the babies' being in "Wakefulness, REM, N-REM / EVRE I, N-REM / EVRE II, N-REM / EVRE III, N-REM / EVRE III, N-REM / EVRE IV" measured by Bispectral Index (BIS) in 5-minute periods within a 24-hour time cycle will be taken from the BIS monitor records and entered into the "Newborn Circadian Rhythm Follow-up Chart" created by the researcher.

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Kucukoglu, Principal Investigator — Selcuk University
Locations (2):
- Turkey (Türkiye) (2):
  - Selcuk University, Konya
  - Kirsehir Ahi Evran University, Kırşehir

IPD SHARING:
Plan to Share IPD: No
It will be shared after the article is published.

REFERENCES:
- [Result] Caba-Flores MD, Ramos-Ligonio A, Camacho-Morales A, Martinez-Valenzuela C, Viveros-Contreras R, Caba M. Breast Milk and the Importance of Chrononutrition. Front Nutr. 2022 May 12;9:867507. doi: 10.3389/fnut.2022.867507. eCollection 2022. PMID 35634367
- [Result] Huang Q, Lai X, Liao J, Tan Y. Effect of non-pharmacological interventions on sleep in preterm infants in the neonatal intensive care unit: A protocol for systematic review and network meta-analysis. Medicine (Baltimore). 2021 Oct 29;100(43):e27587. doi: 10.1097/MD.0000000000027587. PMID 34713833